CLINICAL TRIAL: NCT04150068
Title: A Phase 2/3 Study to Evaluate the Safety and Efficacy of Long-Acting Capsid Inhibitor GS-6207 in Combination With an Optimized Background Regimen in Heavily Treatment Experienced People Living With HIV-1 Infection With Multidrug Resistance
Brief Title: Study to Evaluate the Safety and Efficacy of Lenacapavir (GS-6207) in Combination With an Optimized Background Regimen (OBR) in Heavily Treatment Experienced Participants Living With HIV-1 Infection With Multidrug Resistance
Acronym: CAPELLA
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-200-4625; 2019-003814-16 (EudraCT Number)
Record Dates: First submitted 2019-10-28; First posted 2019-11-04 (Actual); Results first posted 2021-10-20 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — lenacapavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1A: Lenacapavir (Experimental): Participants with HIV-1 ribonucleic acid (RNA) ≥ 400 copies/mL and with a <0.5 log10 HIV-1 RNA decline at Cohort Selection visit compared with screening visit will receive oral lenacapavir (LEN) 600 mg tablet on Days 1 and 2 and 300 mg tablet on Day 8, while continuing their failing regimen in blinded Functional Monotherapy Period (Baseline to Day 14); followed by unblinded Maintenance Period where participants will receive subcutaneous (SC) LEN 927 mg and will initiate an optimized background regimen (OBR) at Day 1 SC Visit (14 days after the first dose of oral LEN).
  Participants will receive their subsequent SC LEN injection at Week 26 Visit (relative to Day 1 SC). Participants will be given an option to receive SC LEN injection at Weeks 52 and 156, while continuing their OBR, until product becomes accessible to participants through an access program or until Gilead elects to discontinue the study in the country.
  Interventions: Drug: Oral Lenacapavir; Drug: Subcutaneous Lenacapavir; Drug: Failing ARV Regimen; Drug: Optimized Background Regimen (OBR)
- Cohort 1B: Placebo to Lenacapavir (Placebo Comparator): Participants with HIV-1 RNA ≥ 400 copies/mL and with a <0.5 log10 HIV-1 RNA decline at the Cohort Selection visit compared with screening visit will receive oral LEN placebo on Days 1, 2, and 8 while continuing their failing regimen in blinded Functional Monotherapy Period (Baseline to Day 14); followed by unblinded Maintenance Period where participants will receive oral LEN 600 mg on Days 15 and 16 and 300 mg on Day 22, and will initiate an OBR on Day 15. At Day 1 SC (14 days after the first dose of oral LEN), participants will receive SC LEN 927 mg while continuing OBR.
  Participants will receive their subsequent SC LEN injection at Week 26 Visit (relative to Day 1 SC). Participants will be given an option to receive SC LEN injection at Weeks 52 and 156, while continuing their OBR, until the product becomes accessible to participants through an access program or until Gilead elects to discontinue study in the country.
  Interventions: Drug: Oral Lenacapavir; Drug: Oral Lenacapavir Placebo; Drug: Subcutaneous Lenacapavir; Drug: Failing ARV Regimen; Drug: Optimized Background Regimen (OBR)
- Cohort 2: Lenacapavir (Experimental): Participants with a ≥ 0.5 log10 copies/mL HIV-1 RNA decline at the Cohort Selection Visit compared with the screening visit or with HIV-1 RNA < 400 copies/mL or if Cohort 1 is fully enrolled will receive oral LEN 600 mg tablet on Days 1 and 2 and 300 mg tablet on Day 8, and will initiate an OBR on Day 1 in Oral Lead-in Period (Baseline to Day 14); followed by Maintenance Period where participants will receive SC LEN 927 mg at Day 1 SC Visit (14 days after the first dose of oral LEN) while continuing their OBR.
  Participants will receive their subsequent SC LEN injection at Week 26 Visit (relative to Day 1 SC). Participants will be given an option to receive SC LEN injection at Weeks 52 and 156, while continuing their OBR, until the product becomes accessible to participants through an access program or until Gilead elects to discontinue the study in the country.
  Interventions: Drug: Oral Lenacapavir; Drug: Subcutaneous Lenacapavir; Drug: Optimized Background Regimen (OBR)

INTERVENTIONS:
Drug: Oral Lenacapavir — Tablets administered without regard to food
  Other Names: Sunlenca®; GS-6207
Drug: Oral Lenacapavir Placebo — Tablets administered without regard to food
  Arms: Cohort 1B: Placebo to Lenacapavir
Drug: Subcutaneous Lenacapavir — Administered in the abdomen via subcutaneous injections
  Other Names: Sunlenca®; GS-6207
Drug: Failing ARV Regimen — Failing antiretroviral (ARV) regimen defined by the lack of efficacy. Any combination of approved and unapproved agents that could potentially be part of the failing regimen.
  Arms: Cohort 1A: Lenacapavir; Cohort 1B: Placebo to Lenacapavir
Drug: Optimized Background Regimen (OBR) — Optimized background regimen as prescribed by the Investigator

SUMMARY:
The primary objective of this study is to evaluate the antiviral activity of lenacapavir (formerly GS-6207) administered as an add-on to a failing regimen (functional monotherapy) in people with human immunodeficiency virus (HIV) (PWH) with multi-drug resistance (MDR).

ELIGIBILITY:
Key Inclusion Criteria:

* Adult aged ≥ 18 years (at all sites) or adolescent aged ≥ 12 and weighing ≥ 35 kg (at sites in North America and Dominican Republic)
* Currently receiving a stable failing ARV regimen for > 8 weeks
* Have HIV-1 RNA ≥ 400 copies/mL at screening
* Have multidrug resistance (resistance to ≥2 agents from ≥3 of the 4 main classes of ARV)
* Have no more than 2 fully active ARV remaining from the 4 main classes that can be effectively combined to form a viable regimen
* Able and willing to receive an OBR together with lenacapavir
* No Hepatitis C virus (HCV) ongoing infection

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2027-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (75):
- United States (35):
  - Ruane Clinical Research Group Inc, Los Angeles, California
  - Mills Clinical Research, Los Angeles, California
  - Eisenhower Health Center at Rimrock, Palm Springs, California
  - One Community Health, Sacramento, California
  - Yale University; School of Medicine, New Haven, Connecticut
  - Washington Health Institute, Washington D.C., District of Columbia
  - Midland Florida Clinical Research Center, LLC, DeLand, Florida
  - Gary J. Richmond, M.D., P.A., Fort Lauderdale, Florida
  - Midway Immunology and Research Center, Ft. Pierce, Florida
  - Floridian Clinical Research, Hialeah, Florida
  - AIDS Healthcare Foundation - South Beach, Miami Beach, Florida
  - Orlando Immunology Center, Orlando, Florida
  - St. Joseph's Hospital Comprehensive Research Institute, Tampa, Florida
  - Triple O Research Institute, P.A., West Palm Beach, Florida
  - Emory Hospital Midtown Infectious Disease Clinic, Atlanta, Georgia
  - Atlanta ID Group, PC, Atlanta, Georgia
  - Chatham County Health Department, Savannah, Georgia
  - Howard Brown Health Center, Chicago, Illinois
  - Northstar Healthcare, Chicago, Illinois
  - Be Well Medical Center, Berkley, Michigan
  - Southampton Healthcare, Inc., St Louis, Missouri
  - New York-Presbyterian/Queens, Flushing, New York
  - North Shore University Hospital/Division of Infectious Diseases, Manhasset, New York
  - Jacobi Medical Center, The Bronx, New York
  - Atrium Health- Infectious Disease Consultants, Charlotte, North Carolina
  - Perelman Center for Advanced Medicine at the Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - 1265 Union Avenue, 8 East, Memphis, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - St Hope Foundation, Bellaire, Texas
  - AIDS Arms, Inc. DBA Prism Health North Texas, Dallas, Texas
  - North Texas Infectious Diseases Consultants, P.A., Dallas, Texas
  - The Crofoot Research Center, INC., Houston, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Clinical Alliance for Research and Education - Infectious Diseases, LLC (CARE-ID), Annandale, Virginia
- Canada (4):
  - Vancouver ID Research and Care Centre Society, Vancouver, British Columbia
  - Maple Leaf Research/Maple Leaf Medical Clinic, Toronto, Ontario
  - Clinique de médecine urbaine du Quartier Latin, Montreal, Quebec
  - The Ottawa Hospital, Ottawa
- Dominican Republic (2):
  - Instituto Dominicano de Estudios Virologicos (IDEV), Santo Domingo
  - Hospital Dr. Salvador Bienvenido Gautier, Santo Domingo
- France (4):
  - Hôpital Sainte-Marguerite, Marseille
  - Hôpital Saint-Louis, Paris
  - Hôpital Saint-Antoine, Paris
  - Hôpital Bichat-Claude Bernard, Paris
- Germany (3):
  - Universitätsklinikum Frankfurt, Medizinische Klinik II, Frankfurt am Main, Hesse
  - Universitätsklinikum Essen, Klinik für Dermatologie und Venerologie, Essen
  - ICH Study Center GmbH & Co. KG, Hamburg
- Italy (5):
  - University of Naples Federico II, Bergamo
  - UOC Malattie Infettive - ASST Spedali Civili Di Brescia - Piazzale Spedali Civili 1, Brescia
  - Divisione di Malattie Infettive, IRCCS Ospedale San Raffaele, Milan
  - U.O.C. IMMUNODEFICIENZE VIRALI - Istituto Nazionale Malattie Infettive Lazzaro Spallanzani IRCCS, Roma
  - U.O.C. Malattie Infettive - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome
- Japan (4):
  - National Hospital Organization Nagoya Medical Center, Nagoya
  - National Hospital Organization Osaka National Hospital, Osaka
  - Tokyo Medical University Hospital, Tokyo
  - Center Hospital of the National Center for Global Health and Medicine, Tokyo
- South Africa (4):
  - Durban International Clinical Research Site, Enhancing Care Foundation, Durban
  - Helen Joseph Hospital, Johannesburg
  - Vx Pharma, Pretoria
  - Perinatal HIV Research Unit (PHRU), Soweto
- Spain (4):
  - Hospital Universitari Germans Trías i Pujol, Badalona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Taiwan (5):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - National Taiwan University Hospital, Taipei
  - Taoyuan General Hospital, Ministry of Health and Welfare, Taoyuan
- Thailand (5):
  - Thai Red Cross AIDS Research Center, Bangkok
  - Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok
  - Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok
  - Faculty of Medicine, Khon Kaen University, Khon Kaen
  - Bamrasnaradura Infectious Diseases Institute, Nonthaburi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Segal-Maurer S, Castagna A, Berhe M, et al. Potent Antiviral Activity of Lenacapavir in Phase 2/3 in Heavily ART-Experienced PWH [Abstract 127]. Presented at: Conference on Retroviruses and Opportunistic Infections; 2021 March 6-10.
- [Derived] Ogbuagu O, Molina JM, Chetchotisakd P, Ramgopal MN, Sanchez W, Brunetta J, Castelli F, Crofoot GE, Hung CC, Ronot-Bregigeon S, Margot NA, Wang H, Dvory-Sobol H, Rhee MS, Segal-Maurer S. Efficacy and Safety of Long-Acting Subcutaneous Lenacapavir in Heavily Treatment-Experienced People with Multidrug-Resistant HIV-1: Week 104 Results of a Phase 2/3 Trial. Clin Infect Dis. 2025 Mar 17;80(3):566-574. doi: 10.1093/cid/ciae423. PMID 39206943
- [Derived] Ogbuagu O, Segal-Maurer S, Ratanasuwan W, Avihingsanon A, Brinson C, Workowski K, Antinori A, Yazdanpanah Y, Trottier B, Wang H, Margot N, Dvory-Sobol H, Rhee MS, Baeten JM, Molina JM; GS-US-200-4625 investigators. Efficacy and safety of the novel capsid inhibitor lenacapavir to treat multidrug-resistant HIV: week 52 results of a phase 2/3 trial. Lancet HIV. 2023 Aug;10(8):e497-e505. doi: 10.1016/S2352-3018(23)00113-3. Epub 2023 Jul 11. PMID 37451297
- [Derived] Segal-Maurer S, DeJesus E, Stellbrink HJ, Castagna A, Richmond GJ, Sinclair GI, Siripassorn K, Ruane PJ, Berhe M, Wang H, Margot NA, Dvory-Sobol H, Hyland RH, Brainard DM, Rhee MS, Baeten JM, Molina JM; CAPELLA Study Investigators. Capsid Inhibition with Lenacapavir in Multidrug-Resistant HIV-1 Infection. N Engl J Med. 2022 May 12;386(19):1793-1803. doi: 10.1056/NEJMoa2115542. PMID 35544387
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=GS-US-200-4625

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Thailand, Italy, Dominican Republic, Spain, France, Canada, Taiwan, South Africa, Japan, and Germany. The first participant was screened on 21 November 2019. Data submitted represent interim analysis performed on data collected by the Primary Completion Date 05 October 2020, and additional data collected after all participants in Cohort 1 completed Week 26 visit.
Pre-assignment Details: 144 participants were screened.
Groups:
- Cohort 1A: Lenacapavir: Participants with human-immunodeficiency virus-1 ribonucleic acid (HIV-1 RNA) ≥ 400 copies/mL and with a <0.5 log10 HIV-1 RNA decline at the Cohort Selection visit compared with screening visit received oral lenacapavir 600 mg tablet on Days 1 and 2 and 300 mg tablet on Day 8, while continuing their failing regimen (previous anti-retroviral [ARV] regimen of any approved and unapproved agents) in blinded Functional Monotherapy Period (Baseline to Day 14); followed by unblinded Maintenance Period where participants received subcutaneous (SC) lenacapavir 927 mg and initiated an optimized background regimen (OBR; as prescribed by the Investigator) at Day 1 SC Visit (14 days after the first dose of oral lenacapavir). Participants received their subsequent SC lenacapavir injection at the Week 26 Visit (relative to Day 1 SC).
  At Week 52 (relative to Day 1 SC), participants will be given an option to receive SC lenacapavir injections every 6 months (26 weeks), while continuing their OBR, until the product became accessible to participants through an access program or until Gilead elected to discontinue the study in the country.
- Cohort 1B: Placebo to Lenacapavir: Participants with HIV-1 RNA ≥ 400 copies/mL and with a <0.5 log10 HIV-1 RNA decline at the Cohort Selection visit compared with screening visit received oral lenacapavir placebo on Days 1, 2, and 8 while continuing their failing regimen (previous ARV regimen of any approved and unapproved agents) in blinded Functional Monotherapy Period (Baseline to Day 14); followed by unblinded Maintenance Period where participants received oral lenacapavir 600 mg tablet on Days 15 and 16 and 300 mg on Day 22, and initiated an OBR (as prescribed by the Investigator) on Day 15. At Day 1 SC (14 days after the first dose of oral lenacapavir), participants received SC lenacapavir 927 mg while continuing their OBR. Participants received their subsequent SC lenacapavir injection at the Week 26 Visit (relative to Day 1 SC).
  At Week 52 (relative to Day 1 SC), participants will be given an option to receive SC lenacapavir injections every 6 months (26 weeks), while continuing their OBR, until the product became accessible to participants through an access program or until Gilead elected to discontinue the study in the country.
- Cohort 2: Lenacapavir: Participants were enrolled in Cohort 2 if Cohort 1 was fully enrolled or if they did not meet the criteria for randomization in Cohort 1 (ie, they had ≥ 0.5 log10 HIV-1 RNA decline compared to the Screening visit and/or HIV-1 RNA < 400 copies/mL at the Cohort Selection visit). Participants received oral lenacapavir 600 mg tablet on Days 1 and 2 and 300 mg tablet on Day 8, and will initiate an OBR on Day 1 in Oral Lead-in Period (Baseline to Day 14); followed by Maintenance Period where participants received SC lenacapavir 927 mg at Day 1 SC Visit (14 days after the first dose of oral lenacapavir) while continuing their OBR. Participants received their subsequent SC lenacapavir injection at the Week 26 Visit (relative to Day 1 SC).
  At Week 52 (relative to Day 1 SC), participants will be given the option to receive SC lenacapavir injections every 6 months (26 weeks), while continuing their OBR, until the product became accessible to participants through an access program or until Gilead elected to discontinue the study in the country.
Period: Functional Mono/Oral Lead-in (14 Days)
Arm/Group | Cohort 1A: Lenacapavir | Cohort 1B: Placebo to Lenacapavir | Cohort 2: Lenacapavir
Started | 24 | 12 | 36
Completed | 24 | 12 | 36
Not Completed | 0 | 0 | 0
Period: Maintenance Period (Week 26 Analysis)
Arm/Group | Cohort 1A: Lenacapavir | Cohort 1B: Placebo to Lenacapavir | Cohort 2: Lenacapavir
Started (Received Day 1 subcutaneous lenacapavir injection.) | 24 | 12 | 36
Completed | 0 | 0 | 0
Not Completed | 24 | 12 | 36
Not completed — Still on study | 24 | 12 | 35
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included participants who were enrolled and received at least 1 dose of study drug.
Groups:
- Cohort 1A: Lenacapavir: Participants with HIV-1 RNA ≥ 400 copies/mL and with a <0.5 log10 HIV-1 RNA decline at the Cohort Selection visit compared with screening visit received oral lenacapavir 600 mg tablet on Days 1 and 2 and 300 mg tablet on Day 8, while continuing their failing regimen (previous ARV regimen of any approved and unapproved agents) in blinded Functional Monotherapy Period (Baseline to Day 14); followed by unblinded Maintenance Period where participants received SC lenacapavir 927 mg and initiated an OBR (as prescribed by the Investigator) at Day 1 SC Visit (14 days after the first dose of oral lenacapavir). Participants received their subsequent SC lenacapavir injection at the Week 26 Visit (relative to Day 1 SC).
  At Week 52 (relative to Day 1 SC), participants will be given an option to receive SC lenacapavir injections every 6 months (26 weeks), while continuing their OBR, until the product became accessible to participants through an access program or until Gilead elected to discontinue the study in the country.
- Total: Total of all reporting groups
Arm/Group | Cohort 1A: Lenacapavir | Cohort 1B: Placebo to Lenacapavir | Cohort 2: Lenacapavir | Total
Number analyzed (Participants) | 24 | 12 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11.3) | 49 (10.9) | 48 (13.7) | 50 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 3 | 8 | 18
  Male | 17 | 9 | 28 | 54
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race information.
  Participants
    Race: Asian | 2 | 1 | 12 | 15
    Race: Black | 10 | 6 | 11 | 27
    Race: White | 12 | 4 | 13 | 29
    Race: Not Permitted | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of ethnicity information
  Participants
    Ethnicity: Hispanic or Latino | 6 | 4 | 5 | 15
    Ethnicity: Not Hispanic or Latino | 18 | 7 | 31 | 56
    Ethnicity: Not Permitted | 0 | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 0 | 0 | 2 | 2
  Dominican Republic | 0 | 1 | 0 | 1
  France | 0 | 1 | 2 | 3
  Italy | 1 | 0 | 6 | 7
  South Africa | 0 | 0 | 1 | 1
  Spain | 1 | 0 | 0 | 1
  Taiwan | 0 | 0 | 1 | 1
  Thailand | 2 | 1 | 8 | 11
  United States | 20 | 9 | 13 | 42
  Japan | 0 | 0 | 2 | 2
  Germany | 0 | 0 | 1 | 1
HIV-1 RNA (log10 copies/mL) [Mean (Standard Deviation); unit: log10 copies/mL] | 3.97 (0.922) | 4.87 (0.393) | 4.06 (1.164) | 4.17 (1.034)
HIV-1 RNA Categories [Count of Participants; unit: Participants]
  ≤ 100000 copies/mL | 23 | 6 | 29 | 58
  > 100000 copies/mL | 1 | 6 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants in Cohort 1 Achieving a Reduction of ≥ 0.5 log10 Copies/mL in Human Immunodeficiency Virus-1 Ribonucleic Acid (HIV-1 RNA) From Baseline to the End of Functional Monotherapy Period
Time Frame: Baseline up to Day 1 SC Visit (14 days after the first dose of oral lencapavir) or Day 15
Population: Full Analysis Set for the Functional Monotherapy Period analysis included participants who were randomized in the Functional Monotherapy Period and received at least 1 dose of blinded study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1A: Lenacapavir | Cohort 1B: Placebo to Lenacapavir
Number analyzed (Participants) | 24 | 12
percentage of participants | 87.5 | 16.7
Statistical Analysis 1: Comparison: Cohort 1A: Lenacapavir vs Cohort 1B: Placebo to Lenacapavir; Test type: Superiority — The difference in percentage between 2 treatment groups was compared using an unconditional exact method using 2 invert 1-sided tests with an alpha level at 0.05 to evaluate superiority; p < 0.0001, Chan & Zhang method — The P value and 95% confidence interval (CI) for the point estimate of treatment difference in proportions was estimated and constructed using the Chan and Zhang method; Percentage Difference = 70.8, 95% CI 2-sided [34.9 to 90.0]

2. Secondary Outcome: Percentage of Participants in Cohort 1 With Plasma HIV-1 RNA < 50 Copies/mL at Week 26 Based on the US FDA-defined Snapshot Algorithm
Description: The percentage of participants in cohort 1 with plasma HIV-1 RNA < 50 copies/mL at Week 26 was analyzed using the United States Food and Drug Administration (US FDA)-defined snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 26 (26 weeks after first dose of subcutaneous lenacapavir)
Population: Full Analysis Set for the All Lenacapavir Analysis included participants who were enrolled into the study and received at least 1 dose of SC lenacapavir.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1A: Lenacapavir | Cohort 1B: Placebo to Lenacapavir
Number analyzed (Participants) | 24 | 12
percentage of participants | 87.5 [67.6 to 97.3] | 66.7 [34.9 to 90.1]

3. Secondary Outcome: Percentage of Participants in Cohort 1 With Plasma HIV-1 RNA < 200 Copies/mL at Week 26 Based on the US FDA-defined Snapshot Algorithm
Description: The percentage of participants in cohort 1 with plasma HIV-1 RNA < 200 copies/mL at Week 26 was analyzed using the US FDA-defined snapshot algorithm, which defines a participant's virologic response status using only the viral load at the predefined time point within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 26 (26 weeks after first dose of subcutaneous lenacapavir)
Population: Participants in the Full Analysis set for the All Lenacapavir Analysis were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1A: Lenacapavir | Cohort 1B: Placebo to Lenacapavir
Number analyzed (Participants) | 24 | 12
percentage of participants | 95.8 [78.9 to 99.9] | 75.0 [42.8 to 94.5]

4. Secondary Outcome: Percentage of Participants in Cohort 1 With Plasma HIV-1 RNA < 50 Copies/mL at Week 52 Based on the US FDA-defined Snapshot Algorithm
Time Frame: Week 52
Reporting Status: Not Posted

5. Secondary Outcome: Percentage of Participants in Cohort 1 With Plasma HIV-1 RNA < 200 Copies/mL at Week 52 Based on the US FDA-defined Snapshot Algorithm
Time Frame: Week 52
Reporting Status: Not Posted

6. Secondary Outcome: Percentage of Participants in Combined Cohorts 1 and 2 With Plasma HIV-1 RNA < 50 Copies/mL From the First Subcutaneous (SC) Dose of Lenacapavir Based on the US FDA-defined Snapshot Algorithm
Time Frame: Week 104
Reporting Status: Not Posted

7. Secondary Outcome: Percentage of Participants in Combined Cohorts 1 and 2 With Plasma HIV-1 RNA < 200 Copies/mL From the First SC Dose of Lenacapavir Based on the US FDA-defined Snapshot Algorithm
Time Frame: Week 104
Reporting Status: Not Posted

8. Secondary Outcome: Percentage of Participants in Combined Cohorts 1 and 2 With Plasma HIV-1 RNA < 50 Copies/mL From the First SC Dose of Lenacapavir Based on the US FDA-defined Snapshot Algorithm
Time Frame: Week 156
Reporting Status: Not Posted

9. Secondary Outcome: Percentage of Participants in Combined Cohorts 1 and 2 With Plasma HIV-1 RNA < 200 Copies/mL From the First SC Dose of Lenacapavir Based on the US FDA-defined Snapshot Algorithm
Time Frame: Week 156
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Enrollment up to Week 26 (26 weeks after first dose of subcutaneous lenacapavir); Adverse Events: First dose date up to Week 26 (26 weeks after first dose of subcutaneous lenacapavir)
Description: All-Cause Mortality: All Enrolled Analysis Set included participants who were randomized into Cohort 1 or enrolled into Cohort 2. Adverse events: Safety Analysis Set included participants who were enrolled and received at least 1 dose of study drug.
Arm/Group | Cohort 1A: Lenacapavir | Cohort 1B: Placebo to Lenacapavir | Cohort 2: Lenacapavir
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/12 | 1/36
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/12 | 2/36
Other Adverse Events (participants affected / at risk) | 20/24 | 11/12 | 30/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1A: Lenacapavir (N=24) | Cohort 1B: Placebo to Lenacapavir (N=12) | Cohort 2: Lenacapavir (N=36)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic mass (Gastrointestinal disorders) | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1A: Lenacapavir (N=24) | Cohort 1B: Placebo to Lenacapavir (N=12) | Cohort 2: Lenacapavir (N=36)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Cerumen impaction (Ear and labyrinth disorders) | 1 | 1 | 0
Ear swelling (Ear and labyrinth disorders) | 0 | 1 | 0
Hypogonadism (Endocrine disorders) | 0 | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 3 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 1
Nausea (Gastrointestinal disorders) | 4 | 1 | 1
Toothache (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 3
Asthenia (General disorders) | 0 | 1 | 2
Fatigue (General disorders) | 3 | 0 | 0
Injection site erythema (General disorders) | 7 | 2 | 10
Injection site induration (General disorders) | 2 | 0 | 7
Injection site nodule (General disorders) | 8 | 4 | 2
Injection site oedema (General disorders) | 1 | 0 | 2
Injection site pain (General disorders) | 7 | 2 | 9
Injection site pruritus (General disorders) | 2 | 0 | 1
Injection site swelling (General disorders) | 9 | 3 | 9
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 2 | 2
Abscess limb (Infections and infestations) | 0 | 1 | 0
Covid-19 (Infections and infestations) | 1 | 0 | 2
Ear infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 2 | 1
Oral herpes (Infections and infestations) | 0 | 2 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0
Tinea versicolour (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 3
Weight decreased (Investigations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 2
Headache (Nervous system disorders) | 2 | 0 | 3
Neuropathy peripheral (Nervous system disorders) | 2 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 2
Sleep disorder (Psychiatric disorders) | 0 | 1 | 1
Glycosuria (Renal and urinary disorders) | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Bullous haemorrhagic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT04150068/Prot_000.pdf
  • Statistical Analysis Plan: Primary Efficacy Endpoint Analysis (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/68/NCT04150068/SAP_002.pdf
  • Statistical Analysis Plan: Week 26 Interim Analysis (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT04150068/SAP_003.pdf